CLINICAL TRIAL: NCT05040893
Title: A Pilot Feasibility Study of a Physiotherapy-based Tailored Intervention for Long COVID.
Brief Title: A Pilot Study of a PhysiOthErapy-based Tailored Intervention for Long COVID (COVID-19)
Acronym: POETIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-0767
Record Dates: First submitted 2021-09-08; First posted 2021-09-10 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Long COVID; Physiotherapy; COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label pilot study investigating the feasibility of the POETIC intervention. POETIC will test a patient-oriented, outpatient physiotherapy intervention tailored to each patient based on their symptoms, functional limitations, and goals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatient Physiotherapy Intervention (Experimental): POETIC will test a patient-oriented, outpatient physiotherapy intervention tailored to each patient based on their symptoms, functional limitations, and goals. The intervention consists of eight one-on-one, supervised sessions delivered over 8 to 10 weeks, approximately one week apart. Each session will be approximately one hour long.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — Interventions will include:
  1. Education and self-management strategies, including the use of wearable activity and real-time heart rate monitors, to safely guide pacing and activity.
  2. Breathing pattern education and retraining (including diaphragmatic, relaxed, and paced breathing exercises).
  3. Return-to-activity exercise programming (e.g., postural, aerobic, and whole-body strengthening exercises).

SUMMARY:
The purpose of this study is to determine the benefits and feasibility of physiotherapy in the recovery of ongoing symptoms after COVID-19 illness. Long COVID Syndrome (Long COVID) is defined by persistent symptoms (including breathlessness, chest pain and fatigue) after COVID-19 illness that continue for more than 12 weeks and cannot be explained by another diagnosis. The goal of this project is to explore physiotherapy as treatment for patients suffering from Long COVID.

DETAILED DESCRIPTION:
The global pandemic caused by Severe Acute Respiratory Syndrome Coronavirus 2 [COVID-19] has resulted in catastrophic loss of life and significant morbidity in survivors. It is now recognized that a significant number of patients have symptoms lasting for weeks to months after initial infection, a clinical entity termed "Long COVID". For many patients, this has led to an unexpectedly long recovery and has negatively impacted health-related quality of life (QOL). Persisting breathlessness, fatigue and exercise limitation were among the most common patient-reported symptoms after COVID-19 infection, affecting approximately 50% of individuals. Given the heterogeneity in the causes of breathlessness post-COVID, there are no specific medications that can be broadly recommended to alleviate dyspnea among these patients. Breathing retraining, combined with supervised exercise, improves QOL and exercise capacity among patients with various chronic lung diseases and is an important potential strategy that could reduce dyspnea and regain physical function among those with Long COVID. The benefits of physiotherapy are recognized in hospitalized, and critically ill patients, and physiotherapy interventions have been studied among hospitalized patients with acute COVID-19 pneumonia. Physiotherapy may also play an instrumental role in the recovery of ambulatory patients with Long COVID, but few data currently exist.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has English language fluency (approximately grade 8-10 reading level) and is able to provide informed consent.
2. Participant is an adult (aged ≥ 18 years).
3. Confirmed diagnosis of COVID-19 via a positive nasopharyngeal or throat swab within the past 12 months.
4. Persistent symptoms lasting ≥12 weeks since the first positive test, including dyspnea (new or increased from baseline as measured by modified Medical Research Council (mMRC) score ≥1).
5. Normal oxygen saturation (greater than 90%) by pulse oximetry at rest on room air.
6. Participant owns a smart phone, tablet, or computer, and has or is willing to create an email address (for links to REDCap and Zoom).

Exclusion Criteria:

1. Abnormal pulmonary function testing (FEV1/FVC ratio <70, total lung capacity <80% predicted, or diffusing capacity <70% predicted).
2. Pre-existing diagnosis chronic lung disease (Interstitial lung disease, COPD, bronchiectasis, or moderate to severe asthma).
3. Pulmonary embolism.
4. Parenchymal abnormalities on chest radiograph, deemed clinically significant by the pulmonologist.
5. Acute or chronic cardiac disease by medical history (myocardial infarction, myocarditis, cardiomyopathy, arrhythmia, moderate or severe valve disease, ventricular dysfunction).
6. Syncope at rest or exertion (which could indicate clinically significant cardiac disease).
7. Pre-existing diagnosis of a post-viral fatigue syndrome, myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) or fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility (patient recruitment and retention rate) | 120 days
  Feasibility will be determined by recruitment of 12 participants within 3 months, retention of >70% of participants and mean completion of >70% of all supervised physiotherapy sessions.

SECONDARY OUTCOMES:
Quality of life (QOL) | 120 days
  The EuroQol-visual analogue scale (EQ-VAS) will be used to measure QOL. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine and 'The worst health you can imagine. The EQ-VAS is the main patient-reported outcome of interest and has an MCID of 8. In addition, the EQ-5D-5L ( 5-level EuroQol-5D)will be used to measure QOL across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents select the level which most closely matches their health state (no problems, slight problems, moderate problems, severe problems or extreme problems). The choices made within each domain relate to a 1-digit number. Combining these digits results in a 5-digit number, which will be converted into a utility weight.
Self-reported functional status | 120 days
  The Post-COVID Functional Scale (PCFS) will be used to measure participant self-reported functional impairment. It covers the full spectrum of functional outcomes, and focuses on limitations in usual activities in five scale grades (0 - 4). Grade 0 reflects the absence of any functional limitation, and upward of grade 1, symptoms, pain or anxiety are present to an increasing degree. Grade 4 reflects severe functional limitations.
Self-efficacy for symptom management | 120 days
  The PROMIS Self-efficacy for Managing Chronic Conditions item bank will be used to measure self-efficacy to manage symptoms and self-efficacy to manage daily activities in both cases, the 4-item short forms). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with higher scores indicating greater severity of depression.
Six-minute walk test | 120 days
  The distance a patient can walk during six minutes.
One-minute sit-to-stand test | 120 days
  The participant will be asked to fully stand and sit back without using their arms and to perform as many repetitions as they safely can within one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Weatherald, MD, MSc, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Peter Lougheed Centre (PLC), University of Calgary, Calgary, Alberta
  - Rockyview General Hospital, University of Calgary, Calgary, Alberta

REFERENCES:
- [Derived] Lo M, Eiriksson L, Hunter S, Twomey R, Skolnik K, Chen J, Afshar EE, Weatherald J, Lim RK. Individually Tailored Physiotherapy in Persons With Respiratory Symptoms Related to Post-Acute Sequelae of COVID-19: A Feasibility Study With Mixed Methods. Health Sci Rep. 2025 Oct 21;8(10):e71367. doi: 10.1002/hsr2.71367. eCollection 2025 Oct. PMID 41132192